CLINICAL TRIAL: NCT02989090
Title: Electronic Patient Notification of Remote Implantable Cardioverter-Defibrillator (ICD) Monitoring Data: Impact of Patient Engagement on Outcomes in the Merlin.Net™ System
Brief Title: Electronic Patient Notification of Remote ICD Data: Impact of Patient Engagement on Outcomes in the Merlin.Net™
Acronym: ePHR-ICD-SJM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Hospital, Indiana (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Michael Mirro, Chief Academic-Research Officer : Parkview Health System, Parkview Hospital, Indiana
Organization: Parkview Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRC13-0113 ePHR-ICD SJM
Record Dates: First submitted 2015-11-18; First posted 2016-12-12 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Implantable Cardioverter-Defibrillator; Health Information Exchange; Electronic Health Records; Patient Participation
Keywords: Patient Engagement; Defibrillators; Health Records, Personal; Patient Portal
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Intervention Group) (Experimental): Receive Detailed ICD Information-electronic: Receive ICD Patient Notification Summary via MyChart Patient Portal Account - Receive training to familiarize yourself with using the ePHR, MyChart Complete baseline, 3 month and 6 months survey
  Interventions: Other: Receive Detailed ICD Information-electronic
- Group B (Intervention Group) (Active Comparator): Receive Detailed ICD Information-paper: Receive ICD Patient Notification Summary via paper Receive training to familiarize yourself with using the ePHR, MyChart Complete baseline, 3 month and 6 months survey
  Interventions: Other: Receive Detailed ICD Information-paper
- Group C (Control Group) (No Intervention): Receives Standard of Care-No Report Complete baseline, 3 month and 6 months survey

INTERVENTIONS:
Other: Receive Detailed ICD Information-electronic — Receive Detailed ICD Information (Patient Notification Summary Report) via an electronic Patient Portal vs control
  Arms: Group A (Intervention Group)
Other: Receive Detailed ICD Information-paper — Receive Detailed ICD Information (Patient Notification Summary Report) via paper vs control
  Arms: Group B (Intervention Group)

SUMMARY:
Remote monitoring of implantable cardioverter-defibrillators (ICDs) for patients has led to efficient, safe, and satisfying analysis of their device and cardiac status; resulting in an overall improvement in the quality of care for such patients. Despite the efficacy of remote monitoring of ICDs and the satisfaction of patients and providers with the process, there is a desire from patients to have access and view ability of the data their ICD is transmitting. However, methods for making ICD device data directly available to the patients are not currently in place. This study aims to elicit the impact of standardized remote monitoring ICD data to patients through an electronic personal health record (ePHR) on patient engagement, healthcare utilization, and patient-provider communication. For this study, patients with an ICD manufactured by St. Jude Medical and that are undergoing remote monitoring through the remote management system, Merlin.net™, will receive a standardized format of their electronic remote monitoring ICD data in MyChart, the ePHR used at Parkview Health. The standard format for the electronic remote monitoring ICD data, as it is delivered to the patient, will be termed the ICD Patient Notification Summary. Additionally, provider attitudes and perceptions regarding the value of the Patient Notification Summary, its impact on clinic workflow, and patient-provider communication will be collected.

DETAILED DESCRIPTION:
Currently, patients receive a letter by postal mail from their physician's office with a statement about their ICD status. The St. Jude Medical ICD data is managed by the Merlin.net™ remote monitoring system and maintained in the database with periodic transfer to the healthcare providers EHR system.

This is the first large study that will evaluate the impact of transferring information from the ICD manufacturer's remote monitoring system directly into a patient's ePHR for the purpose of making select information readily available to patients in the form of a report, called the ICD Patient Notification Summary.

The ICD Patient Notification Summary will be transmitted to the healthcare providers' EHR system (Epic) from Merlin.net™ as part of the data flow pathway to the patients' ePHR (MyChart). This will ensure that the Arrhythmia Diagnostic Center (ADC) clinic and other healthcare providers will be able to view the same information that the patients will receive.

Baseline:

Patients from the intervention group and control groups will answer a baseline survey. The baseline survey will assess socio-demographic characteristics, patient engagement, and patient satisfaction with the current standard of care as well as patient perceptions about receiving remote monitoring ICD data in their ePHR. The survey will be administered either paper-based or online, using a secure online survey program, Survey Monkey. Patient engagement will be assessed using the short form Patient Activation Measure (PAM) survey copyrighted by Insignia Health.

The Patient Activation Measure (PAM) is a validated survey tool developed by Judith Hibbard, PhD, MPH of the University of Oregon, which assesses the degree a patient acts as an active agent in their own health care. PAM is associated with improved health outcomes6.

Follow-up:

Patients will respond to two follow up surveys in approximately 3 months and 6 months from the baseline survey. The follow up surveys will assess patient engagement, patient satisfaction and perceptions with the ICD Patient Notification Summary or current standard of care as well as technology acceptance, depending on the group randomization. Technology acceptance will be assessed using the Technology Acceptance Model as a framework and will explore patient attitudes regarding ease of use, usefulness and intentions to use the ePHR and ICD Patient Notification Summary.

The Technology Acceptance Model is a commonly used model, originally developed by Fred Davis and Richard Bagozzi, which predicts technology acceptance based on the user's perceived usefulness and perceived ease of use of the technology for a specific purpose 7,8.

Data Collection:

Chart review will be performed to collect past and current data regarding patient's socio-demographic characteristics, comorbidities, laboratory and interventions, and healthcare utilization. These data points will help provide background and descriptive information to supplement the other components of the study. ICD-related data and events as well as measurement and classification of clinic calls will be assessed starting six months prior to the study period and continuing throughout the study period. The amount and type of healthcare utilization in relation to cardiac care will be collected. Data related to the use of MyChart will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Physically and mentally capable of providing an informed consent
3. Patient of PPG-Cardiology
4. Implanted with a St. Jude Medical ICD
5. Undergoing remote monitoring by the Merlin.net™ system
6. Ability to read, write and understand English
7. Have access to computer and/or Internet (Group A and B only)
8. Patient has a scheduled ICD download within the study period at the time of enrollment.

Exclusion Criteria:

1. Does not meet inclusion criteria
2. Unable to physically or cognitively carry out the tasks necessary for activating and/or utilizing an ePHR such as; blindness, loss of function of arms, cognitive impairments (per chart review) that would interfere in learning a new task
3. Designated as part of a vulnerable subject population that the investigator or designee identifies to have compromised autonomy related to potential study participation
4. Currently participating in another Parkview study that involves other ePHR use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Patient Engagement evaluated through Patient Activation Measure (PAM) | Baseline, 3 months, and 6 months
  This validated survey instrument will be utilized in the patient survey to evaluate patient engagement.
Change in health outcomes and healthcare utilization | 6 months retrospective and 6 months prospective
  The number of and reason for ER visits, Hospitalization, Office Visits, and Calls to Clinic will be recorded to evaluate patient health outcomes and healthcare utilization before and during the study.

SECONDARY OUTCOMES:
Change in Technology Acceptance evaluated through Technology Acceptance Model (TAM) | Baseline, 3 months, and 6 months
  This validated survey instrument will be utilized in the patient survey to evaluate technology acceptance.
Providers' attitudes and perceptions evaluated through survey | At study conclusion (approximately 1 year post deployment)
  This survey will be utilized to evaluate providers' attitudes and perceptions of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mirro, MD, Principal Investigator — Parkview Health
Locations (1):
- Parkview Health, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guedon-Moreau L, Lacroix D, Sadoul N, Clementy J, Kouakam C, Hermida JS, Aliot E, Boursier M, Bizeau O, Kacet S; ECOST trial Investigators. A randomized study of remote follow-up of implantable cardioverter defibrillators: safety and efficacy report of the ECOST trial. Eur Heart J. 2013 Feb;34(8):605-14. doi: 10.1093/eurheartj/ehs425. Epub 2012 Dec 13. PMID 23242192
- [Background] Landolina M, Perego GB, Lunati M, Curnis A, Guenzati G, Vicentini A, Parati G, Borghi G, Zanaboni P, Valsecchi S, Marzegalli M. Remote monitoring reduces healthcare use and improves quality of care in heart failure patients with implantable defibrillators: the evolution of management strategies of heart failure patients with implantable defibrillators (EVOLVO) study. Circulation. 2012 Jun 19;125(24):2985-92. doi: 10.1161/CIRCULATIONAHA.111.088971. Epub 2012 May 24. PMID 22626743
- [Background] Buntin MB, Jain SH, Blumenthal D. Health information technology: laying the infrastructure for national health reform. Health Aff (Millwood). 2010 Jun;29(6):1214-9. doi: 10.1377/hlthaff.2010.0503. PMID 20530358
- [Background] Carman KL, Dardess P, Maurer M, Sofaer S, Adams K, Bechtel C, Sweeney J. Patient and family engagement: a framework for understanding the elements and developing interventions and policies. Health Aff (Millwood). 2013 Feb;32(2):223-31. doi: 10.1377/hlthaff.2012.1133. PMID 23381514
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939